CLINICAL TRIAL: NCT02869763
Title: Dose-response Effect of Alcohol Ingestion on Steroid Profile: Gender and Ethnic Aspects
Brief Title: Dose-response Effect of Alcohol Ingestion on Steroid Profile
Acronym: PROFETHYL/2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: World Anti-Doping Agency (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, PhD Pharm D, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROFETHYL/2
Record Dates: First submitted 2016-07-28; First posted 2016-08-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Consumption; Healthy
Keywords: Ethanol; Steroid profile; Pharmacokinetics
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 g ethanol (Experimental): 31 mL of Vodka Absolut® diluted in 369 mL of lemon flavored-water (LFW) Fontvella®.
  A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. Administration of ethanol beverage will be controlled: participants will have 5 minutes to drink each glass.
  Interventions: Dietary Supplement: 10 g ethanol
- 20 g ethanol (Experimental): 63 mL of Vodka Absolut® diluted in 337 mL of lemon flavored-water (LFW) Fontvella®.
  A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. Administration of ethanol beverage will be controlled: participants will have 5 minutes to drink each glass.
  Interventions: Dietary Supplement: 20 g ethanol
- Water (Placebo Comparator): 400 mL of lemon flavored-water Fontvella®. A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. The administration will be controlled: participants will have 5 minutes to drink each glass.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: 10 g ethanol — 31 mL of Vodka Absolut® diluted in 369 mL of lemon flavored-water (LFW) Fontvella®.
  A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. Administration of ethanol beverage will be controlled: participants will have 5 minutes to drink each glass.
  Other Names: Vodka Absolut®
  Arms: 10 g ethanol
Dietary Supplement: 20 g ethanol — 63 mL of Vodka Absolut® diluted in 337 mL of lemon flavored-water (LFW) Fontvella®.
  A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. Administration of ethanol beverage will be controlled: participants will have 5 minutes to drink each glass.
  Other Names: Vodka Absolut®
  Arms: 20 g ethanol
Dietary Supplement: Water — 400 mL of lemon flavored-water Fontvella®. A total volume of 400 mL of the drink will be administered, distributed in three 133 mL cool glasses. The administration will be controlled: participants will have 5 minutes to drink each glass.
  Other Names: Lemon flavored-water Fontvella®
  Arms: Water

SUMMARY:
The aim of the clinical trial is to study the intra-individual variation of steroid profile parameters after experimental administration of different doses of ethanol in Caucasian women.

DETAILED DESCRIPTION:
The introduction of the so called 'endocrine module' of the athlete's biological passport needs to consider the numerous reports showing the effect of ethanol ingestion on the steroid profile. A steroid profile would only be useful for longitudinal monitoring and statistical evaluation if it has not been altered by any uncontrolled circumstance, very particularly alcohol consumption.

There is an urgent need to study the perpetuation that alcohol ingestion causes to the individual steroid profile and if possible establish cut-off values for markers of ethanol ingestion granting that the steroid profile determined has not been affected by such ingestion.

Subjects will be genotyped for genetic deletion polymorphism in the uridine diphosphoglucuronosyltransferase family 2 member B17 gene (UGT2B17) related to testosterone glucuronidation regulation.

The objective of the clinical trial is to study the intra-individual variation of steroid profile parameters as a result of the ingestion of different doses of ethanol in Caucasian women (complementing previous studies performed in men).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy women aged 18 to 55 years. Women will enter in studies at the follicular phase of the menstrual cycle, in order to avoid the interference of estrogens.
* Female subjects (if not postmenopausal) possessing regular menstrual cycle between 26 and 32 days and willing to use effective methods of contraception through the study (sexual abstinence, vasectomized partner, sterilization, intrauterine device, double-barrier method).
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* The body mass index (BMI=weigh/height2) will range from 18.5 to 29.9 kg/m2, and the weight from 50 to 100 kg.
* Understanding and accepting the study procedures and signing the informed consent.
* Agreeing to follow a diet free from ethanol in the 72 hours prior to the start of each session and until the end of the study.
* Subjects with social or recreational alcohol consumption, at least 3 standard drinks/week and subjects with experience in several drunkenness.

Exclusion Criteria:

* Not meeting the inclusion criteria.
* History or clinical evidence of alcoholism, drug abuse, or regular use of psychoactive drugs.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* History of psychiatric disorders.
* Women presenting amenorrhea or who suffer from moderate to intense premenstrual syndrome. Female subjects using hormonal contraceptive hormones.
* Smokers of more than 20 cigarettes per day.
* Taking more than 30 g of alcohol a day
* Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Ingestion of vitamin supplements or antioxidants or nonsteroidal anti-inflammatory drugs in the two weeks preceding the study.
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks.
* Subjects with intolerance or adverse reactions to ethanol.
* Subjects who have suffered a hospitalization caused by alcohol intoxication or who have received treatment for drunkenness
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.
* Subjects who follow a vegetarian diet.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline steroid profile | From one day before administration till 24 hours after administration
  24 hours urine will be collected before each experimental session and also up to 24 hours after administration.
Change from baseline Ethyl glucuronide concentrations | From baseline till 24 hours after administration
  Ethyl glucuronide in urine will be measured by Liquid chromatography-mass spectrometry (LC-MS) using deuterated analogs as Internal Standards.
Change from baseline Urine Ethyl sulfate concentrations | From baseline till 24 hours after administration
  Ethyl sulfate in urine will be measured by Liquid chromatography-mass spectrometry (LC-MS) using deuterated analogs as Internal Standards.

SECONDARY OUTCOMES:
Change from baseline alcohol breath air concentrations | From baseline till 6 hours after administration
  Alcohol concentration in breath air will be determined baseline (pre-administration) and up to 6 hours post-administration.
Urine Creatinine concentrations | From one day before administration till 24 hours after administration
  Creatinine will be determined in each urine sample
Change from baseline subjective effects of ethanol | From baseline till 6 hours after administration
  Participants will self-report their experience on a Visual Analogical Scale (VAS): before administration and till 6h post-administration
Number of Participants with Serious and Non-Serious Adverse Events | Through study completion, an average of 1 year
  Collection of adverse effects spontaneously by the participants and/or observed by the investigators.
Change from baseline heart rate | From baseline to 6 hours after administration
  Monitoring heart rate before administration and till 6h post-administration.
Change from baseline oral temperature | From baseline to 6 hours after administration
  Monitoring oral temperature before administration and till 6h post-administration.
Change from baseline blood pressure | From baseline to 6 hours after administration
  Monitoring blood pressure before administration and till 6h post-administration.
Urine pH | From one day before administration till 24 hours after administration
  pH will be determined in each urine sample
Urine specific gravity | From one day before administration till 24 hours after administration
  Specific gravity will be determined in each urine sample
Uridine diphosphoglucuronosyltransferase family 2 member B17 (UGT2B17) deletion genotype | Baseline
  A blood sample for genotyping will be collected. The buffy coat will be stored a -20 degrees celsius (ºC). If deemed necessary for the interpretation of results, DNA will be extracted and evaluated following quantitative multiplex amplification polymerase chain reaction (PCR) for the evaluation of UGT2B17 deletion and copy number variation (CNVs)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre, PhD, Principal Investigator — IMIM-Hospital del Mar Medical Research Institute; José Antonio Pascual, PhD, Study Chair — IMIM-Hospital del Mar Medical Research Institute
Locations (1):
- Parc Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arranz S, Chiva-Blanch G, Valderas-Martinez P, Medina-Remon A, Lamuela-Raventos RM, Estruch R. Wine, beer, alcohol and polyphenols on cardiovascular disease and cancer. Nutrients. 2012 Jul;4(7):759-781. doi: 10.3390/nu4070759. Epub 2012 Jul 10. PMID 22852062
- [Result] Bagnardi V, Zatonski W, Scotti L, La Vecchia C, Corrao G. Does drinking pattern modify the effect of alcohol on the risk of coronary heart disease? Evidence from a meta-analysis. J Epidemiol Community Health. 2008 Jul;62(7):615-9. doi: 10.1136/jech.2007.065607. PMID 18559444
- [Result] Dahl H, Hammarberg A, Franck J, Helander A. Urinary ethyl glucuronide and ethyl sulfate testing for recent drinking in alcohol-dependent outpatients treated with acamprosate or placebo. Alcohol Alcohol. 2011 Sep-Oct;46(5):553-7. doi: 10.1093/alcalc/agr055. Epub 2011 May 26. PMID 21616946
- [Result] Dahl H, Stephanson N, Beck O, Helander A. Comparison of urinary excretion characteristics of ethanol and ethyl glucuronide. J Anal Toxicol. 2002 May-Jun;26(4):201-4. doi: 10.1093/jat/26.4.201. PMID 12054359
- [Result] Jatlow PI, Agro A, Wu R, Nadim H, Toll BA, Ralevski E, Nogueira C, Shi J, Dziura JD, Petrakis IL, O'Malley SS. Ethyl glucuronide and ethyl sulfate assays in clinical trials, interpretation, and limitations: results of a dose ranging alcohol challenge study and 2 clinical trials. Alcohol Clin Exp Res. 2014 Jul;38(7):2056-65. doi: 10.1111/acer.12407. Epub 2014 Apr 28. PMID 24773137
- [Result] Di Castelnuovo A, Costanzo S, Bagnardi V, Donati MB, Iacoviello L, de Gaetano G. Alcohol dosing and total mortality in men and women: an updated meta-analysis of 34 prospective studies. Arch Intern Med. 2006 Dec 11-25;166(22):2437-45. doi: 10.1001/archinte.166.22.2437. PMID 17159008
- [Result] Falk O, Palonek E, Bjorkhem I. Effect of ethanol on the ratio between testosterone and epitestosterone in urine. Clin Chem. 1988 Jul;34(7):1462-4. PMID 3390919
- [Result] Gaedigk A, Twist GP, Leeder JS. CYP2D6, SULT1A1 and UGT2B17 copy number variation: quantitative detection by multiplex PCR. Pharmacogenomics. 2012 Jan;13(1):91-111. doi: 10.2217/pgs.11.135. Epub 2011 Nov 23. PMID 22111604
- [Result] Grosse J, Anielski P, Sachs H, Thieme D. Ethylglucuronide as a potential marker for alcohol-induced elevation of urinary testosterone/epitestosterone ratios. Drug Test Anal. 2009 Nov;1(11-12):526-30. doi: 10.1002/dta.110. PMID 20355168
- [Result] Halter CC, Dresen S, Auwaerter V, Wurst FM, Weinmann W. Kinetics in serum and urinary excretion of ethyl sulfate and ethyl glucuronide after medium dose ethanol intake. Int J Legal Med. 2008 Mar;122(2):123-8. doi: 10.1007/s00414-007-0180-8. Epub 2007 Jun 9. PMID 17558515
- [Result] Jakobsson J, Ekstrom L, Inotsume N, Garle M, Lorentzon M, Ohlsson C, Roh HK, Carlstrom K, Rane A. Large differences in testosterone excretion in Korean and Swedish men are strongly associated with a UDP-glucuronosyl transferase 2B17 polymorphism. J Clin Endocrinol Metab. 2006 Feb;91(2):687-93. doi: 10.1210/jc.2005-1643. Epub 2005 Dec 6. PMID 16332934
- [Result] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Result] Rinaldi S, Peeters PH, Bezemer ID, Dossus L, Biessy C, Sacerdote C, Berrino F, Panico S, Palli D, Tumino R, Khaw KT, Bingham S, Allen NE, Key T, Jensen MK, Overvad K, Olsen A, Tjonneland A, Amiano P, Ardanaz E, Agudo A, Martinez-Garcia C, Quiros JR, Tormo MJ, Nagel G, Linseisen J, Boeing H, Schulz M, Grobbee DE, Bueno-de-Mesquita HB, Koliva M, Kyriazi G, Thrichopoulou A, Boutron-Ruault MC, Clavel-Chapelon F, Ferrari P, Slimani N, Saracci R, Riboli E, Kaaks R. Relationship of alcohol intake and sex steroid concentrations in blood in pre- and post-menopausal women: the European Prospective Investigation into Cancer and Nutrition. Cancer Causes Control. 2006 Oct;17(8):1033-43. doi: 10.1007/s10552-006-0041-7. PMID 16933054
- [Result] Santner SJ, Albertson B, Zhang GY, Zhang GH, Santulli M, Wang C, Demers LM, Shackleton C, Santen RJ. Comparative rates of androgen production and metabolism in Caucasian and Chinese subjects. J Clin Endocrinol Metab. 1998 Jun;83(6):2104-9. doi: 10.1210/jcem.83.6.4898. PMID 9626146
- [Result] Snell LD, Ramchandani VA, Saba L, Herion D, Heilig M, George DT, Pridzun L, Helander A, Schwandt ML, Phillips MJ, Hoffman PL, Tabakoff B; WHO/ISBRA Study on State and Trait Markers of Alcohol Use and Dependence Investigators. The biometric measurement of alcohol consumption. Alcohol Clin Exp Res. 2012 Feb;36(2):332-41. doi: 10.1111/j.1530-0277.2011.01605.x. Epub 2011 Sep 6. PMID 21895709
- [Result] Sottas PE, Saugy M, Saudan C. Endogenous steroid profiling in the athlete biological passport. Endocrinol Metab Clin North Am. 2010 Mar;39(1):59-73, viii-ix. doi: 10.1016/j.ecl.2009.11.003. PMID 20122450
- [Result] Starcevic B, Butch AW. Genetic variations in UDP-glucuronosyl transferase 2B17: implications for testosterone excretion profiling and doping control programs. Clin Chem. 2008 Dec;54(12):1945-7. doi: 10.1373/clinchem.2008.110106. Epub 2008 Oct 16. No abstract available. PMID 18927247
- [Result] Strahm E, Sottas PE, Schweizer C, Saugy M, Dvorak J, Saudan C. Steroid profiles of professional soccer players: an international comparative study. Br J Sports Med. 2009 Dec;43(14):1126-30. doi: 10.1136/bjsm.2008.056242. Epub 2009 Mar 12. PMID 19282302
- [Result] Thieme D, Grosse J, Keller L, Graw M. Urinary concentrations of ethyl glucuronide and ethyl sulfate as thresholds to determine potential ethanol-induced alteration of steroid profiles. Drug Test Anal. 2011 Nov-Dec;3(11-12):851-6. doi: 10.1002/dta.396. PMID 22213685
- [Result] Xu L, Au Yeung SL, Kavikondala S, Leung GM, Schooling CM. Testosterone concentrations in young healthy US versus Chinese men. Am J Hum Biol. 2014 Jan-Feb;26(1):99-102. doi: 10.1002/ajhb.22482. Epub 2013 Nov 19. PMID 24254402